CLINICAL TRIAL: NCT05560100
Title: Development of an Informed Consent Statement Which Communicates the Risk of Adverse Events Associated With Dry Needling Using an Online Nominal Group
Brief Title: Development of an Informed Consent Statement Which Communicates the Risk of Adverse Events Associated With Dry Needling
Acronym: DNICNGT
Status: Completed | Type: Observational
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-173
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Dry Needling
Keywords: informed consent; adverse event; nominal group technique

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients: Must have participated in >= 1 session of dry needling treatment and not be a healthcare provider.
  Interventions: Other: Nominal Group Technique - 2 to 3 hour virtual meeting
- Dry Needling Experts: (1) Must have >= 5 years of clinical practice performing dry needling and at least ONE of the following secondary criteria:
  1. Certification in Dry Needling
  2. Completion of a manual therapy fellowship that included dry needling training
  3. >= 1 total scholarly product (poster presentation, author of a peer-reviewed publication) involving the use of dry needling
  Interventions: Other: Nominal Group Technique - 2 to 3 hour virtual meeting
- Policy Experts: An individual who has a degree in bioethics with at least ONE of the following criteria:
  1. >= 5 years of experience in obtaining informed consent or an advanced graduate degree in bioethics
  2. Has served on ethics related committee in a healthcare institution or healthcare society/professional association
  3. Is or has been a member of a state licensing board
  Interventions: Other: Nominal Group Technique - 2 to 3 hour virtual meeting
- Legal Experts: An individual who is an attorney and who has had training in health law as evidenced by at least ONE of the following criteria:
  1. Evidence of training based on ONE of the follow:
     1. Concentration/Certification in Health Law
     2. L.L.M in health or medical law
     3. SJD in health law
  2. Experience in litigating medical malpractice cases involving failure to obtain informed consent
  3. Published scholarship on informed consent in an academic journal (>= 1)
  Interventions: Other: Nominal Group Technique - 2 to 3 hour virtual meeting

INTERVENTIONS:
Other: Nominal Group Technique - 2 to 3 hour virtual meeting — Participants will be invited to a 2-3 online virtual online meeting with the goal of constructing and defining elements for producing a risk statement for dry needling that can be used for informed consent.

SUMMARY:
As Dry Needling (DN) continues to see increased use in the clinic, there is a need to establish adverse events that could occur as a result of DN intervention. The adverse events are important to consider when an individual needs to make an informed decision regarding their care. It is important to consider how such information should be presented during the informed consent process to improve an individual's ability to make a sound decision regarding their own personal care.

DETAILED DESCRIPTION:
Dry Needling (DN) has been defined by a Task Force organized by the Federation of State Boards of Physical Therapy (FSBPT) as "a skilled intervention performed by a physical therapist using filiform needles to penetrate the skin and/or underlying tissues to affect change in body structures and functions for the evaluation and management of neuromusculoskeletal conditions, pain, movement impairments, and disability". As DN interest continues to expand and studies continue to show the feasibility of applying DN to a wider range of pathological conditions, there is a need to understand the risks related to the use of DN. Understanding the risks associated with DN will allow for improvements in clinical decision making regarding it's application in the clinic.

Enhancing patient choice is a central theme of medical ethics and law. Informed consent (IC) is the legal process used to promote patient autonomy while concepts of shared decision making (SDM) is a widely promoted ethical approach. IC is a means of respecting the autonomous preferences of persons seeking health care or participation in research. Empowerment of the patient is important in healthcare and can lead to improvements in overall quality of patient care and outcomes.

To date, there has been little research conducted that explored the topic of how risks should be presented during the IC process. The purpose of this study will be to utilize expert consensus to establish a risk statement for adverse events associated with DN that an be used during IC.

ELIGIBILITY:
Inclusion Criteria:

Participants must be 18 years old or above and be able to read/write in English Participants must provide informed consent Participants must meet the criteria of one of the previously defined cohort groups used in the study

Dry Needling Experts

(1) Must have >= 5 years of clinical practice performing dry needling and at least ONE of the following secondary criteria:

1. Certification in Dry Needling
2. Completion of a manual therapy fellowship that included dry needling training
3. >= 1 total scholarly product (poster presentation, author of a peer-reviewed publication) involving the use of dry needling

Legal Expert

An individual who is an attorney and who has had training in health law as evidenced by at least ONE of the following criteria:

1. Training in health law as evidenced by ONE of the following:

   1. Concentration/Certification in Health Law
   2. L.L.M in health or medical law
   3. SJD in health law
2. Experience in litigating medical malpractice cases involving failure to obtain informed consent
3. Published scholarship on informed consent in an academic journal (>= 1) Policy Expert

An individual who has a degree in bioethics with at least ONE of the following criteria:

1. >= 5 years of experience in obtaining informed consent or an advanced graduate degree in bioethics
2. Has served on ethics related committee in a healthcare institution or healthcare society/professional association
3. Is or has been a member of a state licensing board

Patient Must have participated in >= 1 session of dry needling treatment and not be a healthcare provider

Exclusion Criteria:

Participants who did not provide informed consent Participants who did not meet the inclusion criteria of one of the four cohort groups defined in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dry Needling Experts, Legal Experts, Policy Experts, and Patients (Defined with inclusion criteria above).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | Up to 2 hours
  Contains questions about the characteristics of the participants
Ranking of Statements | A 2 hour virtual meeting for participants to rank statements
  Participants will rank statements generated during the meeting to determine which statement best meets consensus within the group

CONTACTS AND LOCATIONS:
Overall Officials: Edmund C Ickert, PhD, Principal Investigator — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitney SN, McGuire AL, McCullough LB. A typology of shared decision making, informed consent, and simple consent. Ann Intern Med. 2004 Jan 6;140(1):54-9. doi: 10.7326/0003-4819-140-1-200401060-00012. PMID 14706973
- [Derived] Ickert EC, Griswold D, Learman K, Cook C. Creation of a risk of harms informed consent form for dry needling: A nominal group technique. Musculoskelet Sci Pract. 2023 Aug;66:102778. doi: 10.1016/j.msksp.2023.102778. Epub 2023 May 24. PMID 37290346